CLINICAL TRIAL: NCT03011255
Title: Phase II Study of Radiation Therapy With Peptide Specific CTL Therapy in Treating Patients With Unresectable, Advanced or Recurrent Esophageal Cancer
Brief Title: Combination of Radiation Therapy and Peptide Specific CTL Therapy in Treating Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shixiu Wu (Other)
Responsible Party: Sponsor-Investigator, Shixiu Wu, director of the hospital, Hangzhou Cancer Hospital
Organization: Hangzhou Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH06
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Neoplasms; Esophageal Diseases; Digestive System Diseases
Keywords: Esophageal cancer; Peptide specific CTL; Radiation
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peptide specific CTL arm (Experimental): peptide specific CTL, radiation
  Interventions: Biological: peptide specific CTL

INTERVENTIONS:
Biological: peptide specific CTL — Radiation: RT to 60 Gy, 5 x per week，for 6 weeks Biological: Peptide specific CTL Peptide specific CTL will be administered by intravenous injection on day 28 of radiation.

SUMMARY:
Immunotherapy is now considered to be one of promising approaches for treating cancer. Radiation therapy has been to be a cornerstone treatment for unresectable advanced esophageal cancer. Radiation-induced mutation genes were identified as new sources of tumor associated antigens using exon sequencing and peptide microarray technologies. Epitope peptides for these targets are able to induce peptide specific cytotoxic T lymphocytes (CTL). In this clinical trial, investigators evaluate the efficacy and safety of peptide specific CTL therapy in combination with radiation therapy in treating patients with unresectable, advanced or recurrent esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have unresectable, locally advanced, recurrent disease of esophageal cancer. Histologically confirmed cancer of the esophagus.
2. measurable disease by CT scan
3. ECOG performance status of 0 to 2
4. Expected survival of at least 3months
5. Laboratory values as follow:

   * Absolute neutrophil count (ANC) ≥ 1.5×109
   * White blood cell count ≥ 3×109/L
   * Platelets ≥ 100×109/L
   * Haemoglobin (Hb) ≥ 10g/dL (patients'Hb should be corrected to >10g/dL before treatment)
   * Adequate liver function (within 1 week prior to randomization)
   * Serum bilirubin ≤ 1.5× ULN
   * Alanine aminotransferase/aspartate transaminase (ALT / AST) ≤ 2.5× ULN
   * Alkaline phosphatase (ALP) ≤ 3× ULN
6. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential:Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Active or uncontrolled infection
4. Prior chemotherapy, radiation therapy or immunotherapy
5. Concurrent treatment with steroid or immunosuppressing agent
6. Patient with peptic ulcer disease
7. Other malignancy within 5 years prior to entry into the study, expect for treated non-melanoma skin cancer and cervical carcinoma in situ
8. Disease to the central nervous system
9. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Local control | two years after enrollment
  occurrence of local or regional progression

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 months
  Number of participants with treatment-related adverse events as assessed by Number of participants with treatment-related adverse events as assessed by treatment-related adverse events assessed by CTCAE v4.0
Objective response rate as assessed by RECIST criteria | 3 months
Time to progression | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No